CLINICAL TRIAL: NCT05017402
Title: Higher Dose of Alglucosidase Alpha for Pompe Disease: Long-term Follow-up Study
Brief Title: Higher Dose of Alglucosidase Alpha for Pompe Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-02-019A
Record Dates: First submitted 2021-08-05; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Glycogen Storage Disease Type II
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Alglucosidase Alfa — Standard dose: 20-25 mg/kg every other week; Higher dose: >25 mg/kg every other week.

SUMMARY:
This study is aimed to investigate that whether the higher dose ERT improve safety and clinical outcomes of Pompe disease patients. Also, wish to develop a new therapeutic recommendation and hope that it could improve the long-term outcomes of Pompe diesease patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Pompe disease
2. Currently receiving ERT with regular clinic visits
3. Agree to sign informed consent

Exclusion Criteria:

1. Lost follow-up for clinical visits
2. Allergy to Myozyme
3. Refuse to sign informed consent

Ages: 0 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The observational population included patients of Pompe disease who were diagnosed and treated in our series.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity | For patient older than 3-year-old, first test before study, then every six months, up to 2-years.
  Pulmonary function test (Units: percentage of predictive value)
Peak expiratory flow | For patient older than 3-year-old, first test before study, then every six months, up to 2-years.
  Pulmonary function test (Units: percentage of predictive value)
Polysomnography | For patient older than 6-month-old, first test before study, then every six months, up to 2-years.
  Comprehensive test used to diagnose sleep disorders.

SECONDARY OUTCOMES:
uGLC4 | uGLC4 will be tested before the treatment, then every three months, up to 2-years.
  Urine glucose tetrasaccharide (Units: mmol/mol Creatinine).
CK | CK will be tested before the treatment, then every three months, up to 2-years.
  Blood creatine kinase (Units: units per liter, U/L).
AST | AST will be tested before the treatment, then every three months, up to 2-years.
  Blood aspartate aminotransferase (Units: units per liter, U/L).
ALT | ALT will be tested before the treatment, then every three months, up to 2-years.
  Blood alanine aminotransferase (Units: units per liter, U/L).
Body weight | The body weight will be monitored before the treatment, then every two weeks, up to 2-years.
  Change of body weight (Unit: kilogram, kg)
Body height | The body height will be monitored before the treatment, then every two weeks, up to 2-years.
  Change of body height (Units: centimeter, cm)
Antibody titers | First test will be one month later after first ERT, then every six months, up to 2-years.
  Alglucosidase alfa IgG antibody titer